CLINICAL TRIAL: NCT01914822
Title: The Effect of Ritalin (Methylphenidate Hydrochloride) on Pain and Auditory Sensitivity: an Exploratory Double-blind Randomized Controlled Trial on Healthy Subjects
Brief Title: The Effect Methylphenidate Hydrochloride on Pain and Auditory Sensitivity in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Eisenberg Elon MD, Director, Pain research Unit, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 275-13-RMB; Ritalin version 5 (Other: Rambam Healthcare Campus)
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Pharmacological Action (PA)
Keywords: Ritalin; methylphenidate hydrochloride; experimental pain
MeSH Terms: interventions — Methylphenidate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylphenidate hydrochloride (Experimental): The study will include two sessions which will be conducted at the same time of the day, one week apart from each other. Each session will last approximately 6 hours. In each session subjects will be exposed to baseline experimental pain models and auditory tests. Then they will receive either one MP SR 20 mg tablet or an identical looking placebo.
  Interventions: Drug: methylphenidate hydrochloride
- Sugar pill (Placebo Comparator): The study will include two sessions which will be conducted at the same time of the day, one week apart from each other. Each session will last approximately 6 hours. In each session subjects will be exposed to baseline experimental pain models and auditory tests. Then they will receive either one MP SR 20 mg tablet or an identical looking placebo.
  Interventions: Drug: Sugar pill (placebo)

INTERVENTIONS:
Drug: methylphenidate hydrochloride
  Arms: methylphenidate hydrochloride
Drug: Sugar pill (placebo)
  Arms: Sugar pill

SUMMARY:
1. To examine whether Ritalin has analgesic properties in healthy subjects.
2. To examine if Ritalin analgesic effect is a pain specific phenomenon or a part of a broader, non-specific effect on high mental functions.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between the ages of 20 to 40
* Healthy subjects without known disease and without any chronic pain
* Subjects without known cognitive problems, which can understand the research and its goals
* Subjects who are not taking any medications
* Subjects without hearing problems
* Subjects without attention deficit disorder (ADHD) problems

Exclusion Criteria:

* Subjects who are known to suffer from any disease or any chronic pain
* Subjects taking psychotropic drugs (except Ritalin) or any analgesics
* Subjects who have any contradictions for ritalin administration
* subjects with suspected cognitive disability

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Experimental pain intensity measured on a visual analogue scale (0-100) | 4 hours

SECONDARY OUTCOMES:
effect of Ritalin on auditory sensitivity, measured by the response to different auditory stimulations | 4 hours
pain intensity (NPS 0-100) in response to thermal stimuli and the measures of the auditory tests. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Elon Eisenberg, MD, Principal Investigator — Rambam Helthcare Campus, Haifa, Israel 31096
Locations (1):
- Rambam Healthcare Campus, Haifa, Israel